CLINICAL TRIAL: NCT04122872
Title: GISAR German Interdisciplinary Sarcoma Registry
Acronym: GISAR
Status: Recruiting | Type: Observational
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Other Study IDs: GISAR
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Sarcoma; Sarcoma,Soft Tissue; Sarcoma of Bone; Carcinosarcoma
Keywords: Sarcoma; Soft Tissue Sarcoma; Sarcoma of Bone; Registry
MeSH Terms: conditions — Sarcoma; Osteosarcoma; Carcinosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — formalin-fixed paraffin-embedded tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with bone or soft tissue sarcomas or carcinosarcomas: Adults ≥18 years, verified for bone or soft tissue sarcomas including bone and soft tissue tumors with borderline histological results or with unclear histological dignity (like giant cell tumors of the bone [GCTB], desmoid tumors, atypical lipomatous tumors) as well as carcinosarcomas - independent of kind of therapy and therapy line. Thus, the registry is open for all subtypes of sarcomas and CS.

SUMMARY:
GISAR has an open and modular setup. It is sought to include as many German sarcoma and CS patients (i.e. sarcoma and CS patients treated in Germany) in the registry as possible. A basic data set should be collected on every included patient). In order to adress specific scientific questions, additionally detailed data can be collected in defined patient groups (e.g. effectiveness / adverse effects of systemic therapies in defined situations) within the context of sub-project add-on modules. This data collection can be prospective or retrospective depending on the sub-project

DETAILED DESCRIPTION:
Sarcomas are rare malignant tumors that affect people of all ages. They can be divided into different subtypes yet having more than 80 different forms of soft tissue sarcomas only. In these terms, it is not remarkable that this high number of subtypes is accompanied by various treatment strategies, often representing multimodal treatments.

In addition, in a growing amount of patients tumors are diagnosed, whose malignant cells have histological, cytological, or molecular properties of both epithelial tumors ("carcinoma") and mesenchymal tumors ("sarcoma").

Such "mixed" sarcomatoid/epithelial tumors ("CS") are categorized as carcinoma considering their epithelial origin. But in most cases, CS seem to be more aggressive, than other carcinomas with the same origin; often they are characterized by rapid growth, invasion, disease recurrence and metastases.

Due to the rarity of CS, only limited information is available about their clinical course and best therapeutic approaches. Because of these uncertainties and the sarcoma-component of the tumors, several CS-patients are referred to sarcomacenters. As many experiences with single CS-cases as possible should be collected and evaluated to better understand the different CS-forms.

Due to the complexity of diagnosis and therapy of sarcomas and of CS it is of high relevance to depict the current treatment landscape and the effects and course of different treatment options to illuminate the best option for each specific patient. This is compassed by this registry, as it aims to collect information and data on treatment and outcome of most of future German sarcoma cases along with retrospective data collection to achieve a most comprehensive data set as well as the possibility to identify alterations / trends in the procedures used for sarcoma diagnosis and therapy over time.

ELIGIBILITY:
Inclusion Criteria:

* Histological verified bone or soft tissue sarcomas including bone and soft tissue tumors with borderline histological results or with unclear histological dignity like giant cell tumors of the bone (GCTB), desmoid tumors, atypical lipomatous tumors etc. - independent of therapy form and therapy line - or Histological verified sarcomatoid carcinomas/ carcinosarcomas: tumors with histological, cytological, or molecular properties of both epithelial tumors ("carcinoma") and mesenchymal tumors ("sarcoma") - independent of therapy form and therapy line.
* Signed informed consent form or equivalent (s. chapter 10)
* Age ≥18 years

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults ≥18 years, verified for bone or soft tissue sarcomas including bone and soft tissue tumors with borderline histological results or with unclear histological dignity (like giant cell tumors of the bone [GCTB], desmoid tumors, atypical lipomatous tumors) as well as carcinosarcomas - independent of kind of therapy and therapy line. Thus, the registry is open for all subtypes of sarcomas and CS.
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2018-11-29 (Actual); Primary Completion 2038-01 (Estimated); Study Completion 2038-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of sarcoma preferably specific to the different subtypes | 1 year
  Generation of epidemiological data
Prevalence of sarcoma preferably specific to the different subtypes | 1 year
  Generation of epidemiological data
Prognosis of sarcoma preferably specific to the different subtypes | 1 year
  Generation of epidemiological data

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr, Study Director — Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest
Locations (21):
- Germany (21):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Vivantes Klinikum Berlin-Spandau, Berlin-Spandau
  - Universitätsklinikum Erlangen, Erlangen
  - Klinikum Frankfurt Höchst, Frankfurt
  - Krankenhaus Nordwest KHNW, Frankfurt
  - Uniklinik Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsmedizin Greifswald, Greifswald
  - University Hospital Halle (Saale), Halle
  - Asklepios Klinik St. Georg, Hamburg
  - Uniklinikum Leipzig, Leipzig
  - Universitätsmedizin Mainz, Mainz
  - Chirurgische Universitätsklinik Mannheim, Mannheim
  - Westfälische Wilhelms-Universität Münster, Münster
  - Klinikum Nürnberg, Nuremberg
  - Barmherzige Brüder Regensburg, Regensburg
  - Uniklinikum Regensburg, Regensburg
  - Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared